CLINICAL TRIAL: NCT07259993
Title: Treatment of Knee Osteoarthritis With Stromal Vascular Fraction Cells: 10-Years Follow-up
Brief Title: Knee Osteoarthritis With Stromal Vascular Fraction Cells
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Michael H Carstens (Other)
Collaborators: Wake Forest University (Other); Ministry of Health Nicaragua (Unknown); Hospital Vivian Pellas, Nicaragua (Unknown); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS-DGRS-MABJ-7536-11-13
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SVF cells treatment (Experimental): Intra-articular injection of SVF cells in the injured knee.
  Interventions: Biological: autologous adipose tissue-derived stromal vascular fraction cells

INTERVENTIONS:
Biological: autologous adipose tissue-derived stromal vascular fraction cells — SVF cells via intra-articular injection into knees
  Other Names: SVF

SUMMARY:
This is an interventional study to treat knees osteoarthritis (KOA) with adipose-derived stromal vascular fraction cell components in sixteen subjects with either unilateral or bilateral symptomatic Kellgren Lawence Grade 3 KOA by intra-articular injection of knees. Later, subjects were followed for safety out and potential benefits.

DETAILED DESCRIPTION:
A prospective, open-label interventional study was conducted to assess safety and evidence of clinical response to administration of intra-articular SVF in 16 patients with symptomatic, radiographic Kellgren Lawence grade 3 KOA. Approximately 55.5 million SVF cells were administered via intra-articular injection into each of the 29 knees; asymptomatic knees remained untreated. Subjects were followed for safety out to six months. Potential benefit was measured using the Knee Injury Osteoarthritis Outcome Scores (KOOS) at baseline (pre-treatment), at 3- and 6-months post-treatment, and then subsequently at 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Radiologically documented Kellgren Lawence grade 3 (moderate) KOA;
* Knee pain rated greater than 4/10 on the linear pain scale;
* Previous treatment history with anti-inflammatory medications or corticosteroid injections

Exclusion Criteria:

* Corticosteroid injection within 3 months prior to SVF treatment
* Taking anticoagulants prior to SVF treatment

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-08-27 (Actual); Primary Completion 2025-07-26 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment related adverse events | 6 months follow-up post intervention
  Documentation of adverse events
Osteoarthritis outcome score (KOOS) | Up to 10 years follow-up post SVF treatment
  Changes in KOOS scores

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Escuela Oscar Danilo Rosales Arguello, León, Nicaragua

REFERENCES:
- [Background] Mathiessen A, Conaghan PG. Synovitis in osteoarthritis: current understanding with therapeutic implications. Arthritis Res Ther. 2017 Feb 2;19(1):18. doi: 10.1186/s13075-017-1229-9. PMID 28148295
- [Background] Primorac D, Molnar V, Rod E, Jelec Z, Cukelj F, Matisic V, Vrdoljak T, Hudetz D, Hajsok H, Boric I. Knee Osteoarthritis: A Review of Pathogenesis and State-Of-The-Art Non-Operative Therapeutic Considerations. Genes (Basel). 2020 Jul 26;11(8):854. doi: 10.3390/genes11080854. PMID 32722615
- [Background] Gao F, Mao X, Wu X. Mesenchymal stem cells in osteoarthritis: The need for translation into clinical therapy. Prog Mol Biol Transl Sci. 2023;199:199-225. doi: 10.1016/bs.pmbts.2023.02.006. Epub 2023 Mar 16. PMID 37678972
- [Background] Carstens MH, Garcia N, Mandayam S, Workeneh B, Pastora I, Calderon C, Bertram KA, Correa D. Safety of Stromal Vascular Fraction Cell Therapy for Chronic Kidney Disease of Unknown Cause (Mesoamerican Nephropathy). Stem Cells Transl Med. 2023 Jan 30;12(1):7-16. doi: 10.1093/stcltm/szac080. PMID 36545894
- [Background] Fodor PB, Paulseth SG. Adipose Derived Stromal Cell (ADSC) Injections for Pain Management of Osteoarthritis in the Human Knee Joint. Aesthet Surg J. 2016 Feb;36(2):229-36. doi: 10.1093/asj/sjv135. Epub 2015 Aug 3. PMID 26238455
- [Background] Carstens M, Martinez-Cerrato J, Garcia L, Rivera B, Bertram K. Safety of adipose-derived stromal vascular fraction cells to treat Parkinson's disease. Parkinsonism Relat Disord. 2025 Mar;132:107214. doi: 10.1016/j.parkreldis.2024.107214. Epub 2024 Nov 28. PMID 39658493